CLINICAL TRIAL: NCT05181735
Title: A Randomized Phase I/ II Multicenter Study Evaluating Combination of Luspatercept in LR-MDS Without RS Having Failed or Being Ineligible to ESA
Brief Title: Study Evaluating Combination of Luspatercept in LR-MDS Without RS Having Failed or Being Ineligible to ESA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COMBOLA; 2021-000596-37 (EudraCT Number)
Record Dates: First submitted 2021-12-20; First posted 2022-01-06 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: MDS; Myelodysplastic Syndromes
Keywords: MDS; LR-MDS; Luspatercept; Eprex; ESA
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — luspatercept; Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Luspatercept alone) (Experimental): Patients will receive Luspatercept 1mg/kg (every 3 weeks) with titration up to max of 1.75mg/kg, subcutaneously on day 1 of each 21 day cycle (every three weeks).
  Interventions: Drug: Luspatercept Injection [Reblozyl]
- Arm B (Luspatercept + EPREX) (Experimental): Patients will receive Luspatercept (at the selected dose according to part A) subcutaneously on day 1 of each 21 day cycle (every three weeks) AND Epoetin alfa: At the selected dose (in part A) per week, subcutaneously, every week
  Doses schedules Part A :
  * Level 1 : Luspatercept 0.8 mg/kg + EPREX 30000 UI
  * Level 2 : Luspatercept 1.33 mg/kg + EPREX 30000 UI
  * Level 3 : Luspatercept 1.75mg/kg + EPREX 30000 UI
  * Level 4 : Luspatercept 1.75mg/kg + EPREX 60000 UI
  Interventions: Drug: Luspatercept Injection [Reblozyl]; Drug: Eprex

INTERVENTIONS:
Drug: Luspatercept Injection [Reblozyl] — All patients will receive Luspatercept subcutaneously on day 1 of each 21 day cycle (every 3 weeks) at the selected dose according to part A : 1.75mg/kg or 1.33 mg/kg or 0.8 mg/kg
  Other Names: ACE-536
Drug: Eprex — Epoietin alfa will be adminstered as a subcutaneous injection at the selected dose according to part A : 30 000 UI/week or 60 000 UI/week, every week
  Other Names: Epoietin alfa
  Arms: Arm B (Luspatercept + EPREX)

SUMMARY:
Study of the combination of luspatercept in low-risk myelodysplastic syndrom (LR-MDS) without ring sideroblasts (RS) having failed or being ineligible to ESA

DETAILED DESCRIPTION:
Part A of the trial=Dose-finding Study: Determination the optimal dose level in terms of both toxicity and efficacy for luspatercept + ESA

Part B : Determination of the superiority and efficacy of the association Luspatercept+ESA (erythroipoiesis Stimulating Agent) over luspatercept alone in patients with lower risk MDS who failed to achieve a response or who subsequently relapsed after ESA, wihtout disease progression

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to participate in the study:

* Myelodysplastic syndrome according to current WHO classification
* Age ≥ 18 years
* Patients with lower risk MDS according to IPSS classification (LOW, INT-1) without RS who failed to achieved a response or who subsequently relapse after ESA (at least 60000 U EPO-a over at least 12weeks or equivalent), without disease progression (or ineligible to ESA defined by EPO > 500 UI/l)
* Hemoglobin < 9 gr/dl or Transfusion dependant (at least 3 RBCs in 16 wk in at least 2 transfusion episodes)
* Non del(5q) syndrome
* Adequat renal function, defined by creatinine less than 1.5 times the upper limit of normal, creatinine clearance ≥ 40 mL/min (MDRD formula).
* Adequat liver function, defined by total bilirubin and transaminases less than 1.5 times the upper limit of normal.
* Patient is not known to be refractory to platelet transfusions.
* Written informed consent.
* Patient must understand and voluntarily sign consent form.
* Patient must be able to adhere to the visit schedule as outlined in the study and follow protocol requirements.
* ECOG performance status 0-2 at the time of screening.
* A FCBP (female of childbearing potential) for this study was defined as a sexually mature woman who: (1) had not undergone a hysterectomy or bilateral oophorectomy; or (2) had not been naturally postmenopausal (amenorrhea following cancer therapy did not rule out childbearing potential) for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months). A FCBP participating in the study must:

  * Have had 2 negative pregnancy tests as verified by the investigator prior to starting IP (unless the screening pregnancy test was done within 72 hours of Cycle 1 Day 1). She must have had agreed to ongoing a monthly pregnancy testing during the course of the study and after EOT
  * If sexually active, agreed to have used, and been able to comply with, highly effective contraception** without interruption, 5 weeks prior to starting IP, during treatment with IP (including dose interruptions), and for 12 weeks after discontinuation of IP.
  * ** Highly effective contraception was defined in this protocol as the following (information also appeared in the ICF): Hormonal contraception (eg, birth control pills, injection, implant, transdermal patch, vaginal ring), intrauterine device, tubal ligation (tying your tubes), or a partner with a vasectomy
* Male subjects must: Have agreed to use a condom, defined as a male latex condom or nonlatex condom NOT made out of natural (animal) membrane (eg, polyurethane), during sexual contact with a pregnant female or a FCBP while participating in the study, during dose interruptions, and for at least 12 weeks following IP discontinuation, even if he had undergone a successful vasectomy

Exclusion Criteria:

A patient meeting any of the following criteria is not eligible to participate in the study:

* Severe infection or any other uncontrolled severe condition.
* Uncontrolled hypertension
* Significant cardiac disease - NYHA Class III or IV or having suffered a myocardial infarction in the last 6 months.
* del(5q) syndrome
* Use of investigational agents within 30 days or any anticancer therapy (including IMiD) within 2 weeks before the study entry with the exception of hydroxyurea. The patient must have recovered at least a grade 1 from all acute toxicity from any previous therapy.
* Use of EPO within 4 weeks before the study entry
* Active cancer, or cancer during the year prior to trial entry other than basal cell carcinoma, or carcinoma in situ of the cervix or breast.
* Patient already enrolled in another therapeutic trial of an investigational drug.
* Known HIV infection or active hepatitis B or C.
* Women who are or could become pregnant or who are currently breastfeeding.
* Any medical or psychiatric contraindication that would prevent the patient from understanding and signing the informed consent form.
* Patient eligible for allogeneic stem cell transplantation.
* Known allergies to luspatercept or EPO or any of its excipients.
* No affiliation to a health insurance system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2028-12-19 (Estimated); Study Completion 2029-06-19 (Estimated)

PRIMARY OUTCOMES:
Part A : Dose-finding study | Evaluation of Dose-limiting toxicity (DLT) at Day 21 of cycle 1 for non-hematological toxicity , up to day 42 for hematological toxicity
  To determine the optimal dose level in terms of both toxicity and efficacy for luspatercept + EPO
Part B : Benefit of the association over the monotherapy | At week 25
  To determine, at Week 25, the superiority and efficacy of luspatercept + ESA over luspatecept alone

SECONDARY OUTCOMES:
Response rate | 3 months
  To determine the response rate (complete response (CR) +Partial Response (PR) + stable disease with Hematological Improvment (HI) according to IWG 2006 criteria) in each arm
Response duration | 24 months
  Duration of response ends with date loss of response, relapse or death whichever occurs first
Overall survival | 30 months
  Overall survival time ends for patients who die during the follow up period with the date of death and for patients who do not die during the follow up period with the date when the patient was last seen to be alive

CONTACTS AND LOCATIONS:
Overall Officials: Lionel ADES, Pr., Principal Investigator — Hôpital Saint Louis
Locations (38):
- France (38):
  - CHU Amiens-Picardie, Amiens
  - Clinique de l'Europe, Amiens
  - CHU Angers, Angers
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - CH Henri Duffaut d'Avignon, Avignon
  - Centre Hospitalier de la Côte Basque, Bayonne
  - Hôpital Avicenne, Bobigny
  - Hôpital Privé Sévigné, Cesson-Sévigné
  - CHU de Grenoble, Grenoble
  - Centre Hospitalier de Versailles, Le Chesnay
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CH Le Mans, Le Mans
  - CHRU de Lille - Hôpital Claude Huriez, Lille
  - CHRU de Limoges - Hôpital Dupuytren, Limoges
  - Centre Hospitalier de Mont de Marsan, Mont-de-Marsan
  - CHU Saint Eloi, Montpellier
  - CHU Nantes - Hôtel Dieu, Nantes
  - Hôpital privé du Confluent, Nantes
  - CHU de Nice - Hôpital Archet 1, Nice
  - CHU de Nîmes, Nîmes
  - CHR d'Orléans, Orléans
  - Hôpital Saint Louis, Paris
  - Hôpital Cochin, Paris
  - Hôpital Necker, Paris
  - CHU de Bordeaux - Hôpital Haut-Lévêque, Pessac
  - Centre Hospitalier de Périgueux, Périgueux
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Poitiers, Poitiers
  - Hôpital NOVO, Pontoise
  - Centre Hospitalier de Cornouaille, Quimper
  - CHU de Rennes - Hôpital Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut de Cancérologie et d'Hématologie Universitaire de Saint-Etienne, Saint-Priest-en-Jarez
  - Strasbourg Oncologie Libérale Clinique Sainte Anne, Strasbourg
  - CHU Toulouse - IUCT Oncopole, Toulouse
  - CHU de Tours - Hôpital Bretonneau, Tours
  - Centre Hospitalier de Valence, Valence
  - CHRU Nancy - Hôpitaux de Brabois, Vandœuvre-lès-Nancy